CLINICAL TRIAL: NCT07188246
Title: A Trial of Neoadjuvant, Hypofractionated Radiation, With Intratumoural Pembrolizumab Followed by Neoadjuvant Chemotherapy, in Stage 3 or High-risk Stage 2 Breast Cancer
Brief Title: Neoadjuvant, SBRT With Intratumoural Pembrolizumab Followed by Neoadjuvant Chemotherapy in Breast Cancer
Acronym: BRINK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Muriel Brackstone, Chair/Chief of General Surgery, General Surgeon, Surgical Oncologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 122109
Record Dates: First submitted 2023-05-04; First posted 2025-09-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer Invasive; Breast Cancer Triple Negative
Keywords: Immunotherapy; Pembrolizumab; Breast SBRT
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Radiation; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Single arm open-label study of breast SBRT with immunotherapy before neoadjuvant chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT with Pembrolizumab (Experimental): Stereotactic body radiation therapy delivered to the main breast tumour with 2 injections of pembrolizumab (Keytruda), completed prior to neoadjuvant chemotherapy.
  Interventions: Radiation: Radiation; Drug: Pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Radiation: Radiation — Stereotactic body radiation therapy to the breast
Drug: Pembrolizumab (KEYTRUDA®) — Two injections

SUMMARY:
This study will evaluate the immune-priming effects of stereotactic body radiation therapy (SBRT) regimen coupled with two injections of pembrolizumab in high-risk primary breast carcinoma prior to neoadjuvant chemotherapy. Preliminary results from the investigators' local TRIO Trial suggest that SBRT prior to neoadjuvant chemotherapy (NAC) may result in improved response rates due to the combined effect of radiation therapy (RT) and chemotherapy. The investigators aim to augment this effect with the addition of pembrolizumab, a monoclonal antibody that binds to and blocks programmed cell death protein 1 (PD-1).

DETAILED DESCRIPTION:
This study will evaluate the immune-priming effects of stereotactic body radiation therapy (SBRT) combined with intratumoural pembrolizumab in patients with high-risk primary breast carcinoma prior to neoadjuvant chemotherapy. Prior feasibility trials (SIGNAL and TRIO) demonstrated that neoadjuvant SBRT can upregulate immune-related genes, suggesting conversion of tumors toward an "immune hot" phenotype that may enhance responsiveness to immunotherapy.

The current trial builds on this work by adding pembrolizumab, an anti-PD-1 antibody, to determine whether further immune priming can be achieved. Study objectives include assessing feasibility, safety, molecular immune activation, and preliminary clinical outcomes of this regimen before standard chemotherapy.

SBRT is a highly targeted radiotherapy technique that has demonstrated feasibility in early and locally advanced breast cancer trials, with low toxicity. Pembrolizumab is approved for multiple cancers, including triple negative breast cancer, and may act synergistically with radiotherapy to enhance antitumor immune responses. Findings from this study will inform future randomized trials evaluating whether combining SBRT and immunotherapy can improve pathologic complete response rates and long-term outcomes in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive ductal carcinoma of any subtype (including invasive mammary carcinoma with lobular features), excluding sarcomatous, signet or metaplastic subtypes.
2. Invasive mammary carcinoma of stages IIB - III (excluding inflammatory breast cancer). Stage IIA is eligible for triple negative and HER2+ breast cancers.

   a. Clinical staging based on AJCC 8th edition.
3. Lesion palpable by treating physician.
4. Plan to be treated with neoadjuvant chemotherapy.
5. Able to tolerate core needle biopsies and pembrolizumab injection.
6. 18 years of age or older.
7. Able to provide informed consent.

Exclusion Criteria:

1. Any serious medical comorbidities or other contraindications to radiotherapy, chemotherapy, or surgery (e.g., uncontrolled diabetes, serious heart condition, etc).
2. Prior treatment for current breast cancer.
3. Previous radiation therapy to the same breast.
4. Inflammatory breast carcinoma.
5. Invasive mammary carcinoma with sarcomatous, signet cell or metaplastic subtypes.
6. Recurrent breast cancer.
7. Clinical or radiologic evidence or suspicion of distant metastatic disease (metastatic workup that requires additional imaging to follow-up on suspicious findings will exclude patients).
8. Any collagen vascular disease precluding radiotherapy at the discretion of the treating radiation oncologist (particularly lupus, scleroderma, dermatomyositis, psoriatic arthritis).
9. No prior stem cell transplantation.
10. Any poorly controlled autoimmune conditions.
11. Current use of corticosteroids or immunosuppressants.
12. Any other malignancy at any site (except non-melanomatous skin cancer) <5 years prior to study enrollment. Synchronous bilateral breast cancers are acceptable.
13. Inability to tolerate core needle biopsies or pembrolizumab injection.
14. Pregnant or lactating.
15. Under 18 years of age.
16. Inability or unwillingness to provide informed consent.
17. Inability or unwillingness to complete study assessments/interventions and follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response | Measured at time of surgery, typically 6 months after enrollment in trial.
  Pathologic complete response rates after neoadjuvant radiotherapy, pembrolizumab and chemotherapy will be evaluated.

SECONDARY OUTCOMES:
Immune priming | Measured 3 to 8 days after last dose of pembrolizumab. Which is Day 20-25, where blood and tissue will be collected.
  To evaluate the degree of immune priming in this regimen compared descriptively to TRIO Trial
Breast and skin tissue adverse events to evaluate toxicity of treatment | Baseline, 3 weeks post-op, 6 months post-op, 1 year post-op
  Toxicity to surrounding breast and skin tissue, defined by ≥ grade 2 fibrosis.
Treatment related adverse event | Measured at up to surgery, typically 6 months after enrolment in trial.
  Adverse events relating to the interventional radiation or pembrolizumab defined by ≥ grade 3
Local Recurrence Rates | Disease status will be evaluated at routine patient follow-up appointments, including yearly mammography. Will be recorded at Year 1, Year 2, Year 3, Year 4, Year 5
  Ipsilateral breast recurrence rate.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barendsen GW. Dose fractionation, dose rate and iso-effect relationships for normal tissue responses. Int J Radiat Oncol Biol Phys. 1982 Nov;8(11):1981-97. doi: 10.1016/0360-3016(82)90459-x. No abstract available. PMID 6759484
- [Background] Beal K, McCormick B, Zelefsky MJ, Borgen P, Fey J, Goldberg J, Cohen GN, Sacchini V. Single-fraction intraoperative radiotherapy for breast cancer: early cosmetic results. Int J Radiat Oncol Biol Phys. 2007 Sep 1;69(1):19-24. doi: 10.1016/j.ijrobp.2007.02.010. Epub 2007 Apr 18. PMID 17446003
- [Background] Blitzblau RC, Arya R, Yoo S, Baker JA, Chang Z, Palta M, Duffy E, Horton JK. A phase 1 trial of preoperative partial breast radiation therapy: Patient selection, target delineation, and dose delivery. Pract Radiat Oncol. 2015 Sep-Oct;5(5):e513-e520. doi: 10.1016/j.prro.2015.02.002. Epub 2015 Mar 31. PMID 25834942
- [Background] Bondiau PY, Courdi A, Bahadoran P, Chamorey E, Queille-Roussel C, Lallement M, Birtwisle-Peyrottes I, Chapellier C, Pacquelet-Cheli S, Ferrero JM. Phase 1 clinical trial of stereotactic body radiation therapy concomitant with neoadjuvant chemotherapy for breast cancer. Int J Radiat Oncol Biol Phys. 2013 Apr 1;85(5):1193-9. doi: 10.1016/j.ijrobp.2012.10.034. Epub 2013 Jan 16. PMID 23332384
- [Background] Cortes J, Cescon DW, Rugo HS, Nowecki Z, Im SA, Yusof MM, Gallardo C, Lipatov O, Barrios CH, Holgado E, Iwata H, Masuda N, Otero MT, Gokmen E, Loi S, Guo Z, Zhao J, Aktan G, Karantza V, Schmid P; KEYNOTE-355 Investigators. Pembrolizumab plus chemotherapy versus placebo plus chemotherapy for previously untreated locally recurrent inoperable or metastatic triple-negative breast cancer (KEYNOTE-355): a randomised, placebo-controlled, double-blind, phase 3 clinical trial. Lancet. 2020 Dec 5;396(10265):1817-1828. doi: 10.1016/S0140-6736(20)32531-9. PMID 33278935
- [Background] Cortes J, Rugo HS, Cescon DW, Im SA, Yusof MM, Gallardo C, Lipatov O, Barrios CH, Perez-Garcia J, Iwata H, Masuda N, Torregroza Otero M, Gokmen E, Loi S, Guo Z, Zhou X, Karantza V, Pan W, Schmid P; KEYNOTE-355 Investigators. Pembrolizumab plus Chemotherapy in Advanced Triple-Negative Breast Cancer. N Engl J Med. 2022 Jul 21;387(3):217-226. doi: 10.1056/NEJMoa2202809. PMID 35857659
- [Background] Dai M, Yip YY, Hellstrom I, Hellstrom KE. Curing mice with large tumors by locally delivering combinations of immunomodulatory antibodies. Clin Cancer Res. 2015 Mar 1;21(5):1127-38. doi: 10.1158/1078-0432.CCR-14-1339. Epub 2014 Aug 20. PMID 25142145
- [Background] Demaria S, Romano E, Brackstone M, Formenti SC. Immune induction strategies to enhance responses to PD-1 blockade: lessons from the TONIC trial. J Immunother Cancer. 2019 Nov 21;7(1):318. doi: 10.1186/s40425-019-0783-x. PMID 31752991
- [Background] Dewan MZ, Galloway AE, Kawashima N, Dewyngaert JK, Babb JS, Formenti SC, Demaria S. Fractionated but not single-dose radiotherapy induces an immune-mediated abscopal effect when combined with anti-CTLA-4 antibody. Clin Cancer Res. 2009 Sep 1;15(17):5379-88. doi: 10.1158/1078-0432.CCR-09-0265. Epub 2009 Aug 25. PMID 19706802
- [Background] Dunlap NE, Cai J, Biedermann GB, Yang W, Benedict SH, Sheng K, Schefter TE, Kavanagh BD, Larner JM. Chest wall volume receiving >30 Gy predicts risk of severe pain and/or rib fracture after lung stereotactic body radiotherapy. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):796-801. doi: 10.1016/j.ijrobp.2009.02.027. Epub 2009 May 8. PMID 19427740
- [Background] Eaton DJ, Best B, Brew-Graves C, Duck S, Ghaus T, Gonzalez R, Pigott K, Reynolds C, Williams NR, Keshtgar MR. In vivo dosimetry for single-fraction targeted intraoperative radiotherapy (TARGIT) for breast cancer. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):e819-24. doi: 10.1016/j.ijrobp.2011.11.012. Epub 2012 Jan 31. PMID 22300571
- [Background] Edwards AA, Keggin E, Plowman PN. The developing role for intensity-modulated radiation therapy (IMRT) in the non-surgical treatment of brain metastases. Br J Radiol. 2010 Feb;83(986):133-6. doi: 10.1259/bjr/28596848. Epub 2009 Dec 17. PMID 20019176
- [Background] Glencer AC, Wong JM, Hylton NM, Krings G, McCune E, Rothschild HT, Loveday TA, Alvarado MD, Esserman LJ, Campbell MJ. Modulation of the immune microenvironment of high-risk ductal carcinoma in situ by intralesional pembrolizumab injection. NPJ Breast Cancer. 2021 May 25;7(1):59. doi: 10.1038/s41523-021-00267-z. PMID 34035311
- [Background] Greco C, Zelefsky MJ, Lovelock M, Fuks Z, Hunt M, Rosenzweig K, Zatcky J, Kim B, Yamada Y. Predictors of local control after single-dose stereotactic image-guided intensity-modulated radiotherapy for extracranial metastases. Int J Radiat Oncol Biol Phys. 2011 Mar 15;79(4):1151-7. doi: 10.1016/j.ijrobp.2009.12.038. Epub 2010 May 25. PMID 20510537
- [Background] Hong WX, Haebe S, Lee AS, Westphalen CB, Norton JA, Jiang W, Levy R. Intratumoral Immunotherapy for Early-stage Solid Tumors. Clin Cancer Res. 2020 Jul 1;26(13):3091-3099. doi: 10.1158/1078-0432.CCR-19-3642. Epub 2020 Feb 18. PMID 32071116
- [Background] Hoppe BS, Laser B, Kowalski AV, Fontenla SC, Pena-Greenberg E, Yorke ED, Lovelock DM, Hunt MA, Rosenzweig KE. Acute skin toxicity following stereotactic body radiation therapy for stage I non-small-cell lung cancer: who's at risk? Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1283-6. doi: 10.1016/j.ijrobp.2008.08.036. PMID 19028267
- [Background] Iaccarino G, Pinnaro P, Landoni V, Marzi S, Soriani A, Giordano C, Arcangeli S, Benassi M, Arcangeli G. Single fraction partial breast irradiation in prone position. J Exp Clin Cancer Res. 2007 Dec;26(4):543-52. PMID 18365551
- [Background] Keshtgar MR, Vaidya JS, Tobias JS, Wenz F, Joseph D, Stacey C, Metaxas MG, Keller A, Corica T, Williams NR, Baum M. Targeted intraoperative radiotherapy for breast cancer in patients in whom external beam radiation is not possible. Int J Radiat Oncol Biol Phys. 2011 May 1;80(1):31-8. doi: 10.1016/j.ijrobp.2010.01.045. Epub 2010 Jun 18. PMID 20646864
- [Background] Kimple RJ, Klauber-DeMore N, Kuzmiak CM, Pavic D, Lian J, Livasy CA, Chiu WM, Moore DT, Sartor CI, Ollila DW. Local control following single-dose intraoperative radiotherapy prior to surgical excision of early-stage breast cancer. Ann Surg Oncol. 2011 Apr;18(4):939-45. doi: 10.1245/s10434-010-1392-6. PMID 21061074
- [Background] Lemanski C, Azria D, Gourgon-Bourgade S, Gutowski M, Rouanet P, Saint-Aubert B, Ailleres N, Fenoglietto P, Dubois JB. Intraoperative radiotherapy in early-stage breast cancer: results of the montpellier phase II trial. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):698-703. doi: 10.1016/j.ijrobp.2009.02.039. Epub 2009 May 23. PMID 19467579
- [Background] Marabelle A, Kohrt H, Sagiv-Barfi I, Ajami B, Axtell RC, Zhou G, Rajapaksa R, Green MR, Torchia J, Brody J, Luong R, Rosenblum MD, Steinman L, Levitsky HI, Tse V, Levy R. Depleting tumor-specific Tregs at a single site eradicates disseminated tumors. J Clin Invest. 2013 Jun;123(6):2447-63. doi: 10.1172/JCI64859. PMID 23728179
- [Background] Melero I, Castanon E, Alvarez M, Champiat S, Marabelle A. Intratumoural administration and tumour tissue targeting of cancer immunotherapies. Nat Rev Clin Oncol. 2021 Sep;18(9):558-576. doi: 10.1038/s41571-021-00507-y. Epub 2021 May 18. PMID 34006998
- [Background] Middleton MR, Hoeller C, Michielin O, Robert C, Caramella C, Ohrling K, Hauschild A. Intratumoural immunotherapies for unresectable and metastatic melanoma: current status and future perspectives. Br J Cancer. 2020 Sep;123(6):885-897. doi: 10.1038/s41416-020-0994-4. Epub 2020 Jul 27. PMID 32713938
- [Background] Minniti G, Salvati M, Muni R, Lanzetta G, Osti MF, Clarke E, Costa A, Bozzao A, Trasimeni G, Enrici RM. Stereotactic radiosurgery plus whole-brain radiotherapy for treatment of multiple metastases from non-small cell lung cancer. Anticancer Res. 2010 Jul;30(7):3055-61. PMID 20683055
- [Background] Ollila DW, Klauber-DeMore N, Tesche LJ, Kuzmiak CM, Pavic D, Goyal LK, Lian J, Chang S, Livasy CA, Sherron RF, Sartor CI. Feasibility of breast preserving therapy with single fraction in situ radiotherapy delivered intraoperatively. Ann Surg Oncol. 2007 Feb;14(2):660-9. doi: 10.1245/s10434-006-9154-1. PMID 17091330
- [Background] Palma D, Visser O, Lagerwaard FJ, Belderbos J, Slotman BJ, Senan S. Impact of introducing stereotactic lung radiotherapy for elderly patients with stage I non-small-cell lung cancer: a population-based time-trend analysis. J Clin Oncol. 2010 Dec 10;28(35):5153-9. doi: 10.1200/JCO.2010.30.0731. Epub 2010 Nov 1. PMID 21041709
- [Background] Palta M, Yoo S, Adamson JD, Prosnitz LR, Horton JK. Preoperative single fraction partial breast radiotherapy for early-stage breast cancer. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):37-42. doi: 10.1016/j.ijrobp.2010.09.041. Epub 2010 Nov 17. PMID 21093166
- [Background] Park C, Papiez L, Zhang S, Story M, Timmerman RD. Universal survival curve and single fraction equivalent dose: useful tools in understanding potency of ablative radiotherapy. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):847-52. doi: 10.1016/j.ijrobp.2007.10.059. PMID 18262098
- [Background] Pinnaro P, Arcangeli S, Giordano C, Arcangeli G, Impiombato FA, Pinzi V, Iaccarino G, Soriani A, Landoni V, Strigari L. Toxicity and cosmesis outcomes after single fraction partial breast irradiation in early stage breast cancer. Radiat Oncol. 2011 Nov 11;6:155. doi: 10.1186/1748-717X-6-155. PMID 22079051
- [Background] Sacchini V, Beal K, Goldberg J, Montgomery L, Port E, McCormick B. Study of quadrant high-dose intraoperative radiation therapy for early-stage breast cancer. Br J Surg. 2008 Sep;95(9):1105-10. doi: 10.1002/bjs.6208. PMID 18690634
- [Background] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- [Background] Theberge V, Whelan T, Shaitelman SF, Vicini FA. Altered fractionation: rationale and justification for whole and partial breast hypofractionated radiotherapy. Semin Radiat Oncol. 2011 Jan;21(1):55-65. doi: 10.1016/j.semradonc.2010.08.007. PMID 21134655
- [Background] Vaidya JS, Baum M, Tobias JS, Wenz F, Massarut S, Keshtgar M, Hilaris B, Saunders C, Williams NR, Brew-Graves C, Corica T, Roncadin M, Kraus-Tiefenbacher U, Sutterlin M, Bulsara M, Joseph D. Long-term results of targeted intraoperative radiotherapy (Targit) boost during breast-conserving surgery. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):1091-7. doi: 10.1016/j.ijrobp.2010.07.1996. Epub 2010 Oct 15. PMID 20951505
- [Background] Vaidya JS, Hall-Craggs M, Baum M, Tobias JS, Falzon M, D'Souza DP, Morgan S. Percutaneous minimally invasive stereotactic primary radiotherapy for breast cancer. Lancet Oncol. 2002 Apr;3(4):252-3. doi: 10.1016/s1470-2045(02)00717-9. No abstract available. PMID 12067688
- [Background] Vaidya JS, Joseph DJ, Tobias JS, Bulsara M, Wenz F, Saunders C, Alvarado M, Flyger HL, Massarut S, Eiermann W, Keshtgar M, Dewar J, Kraus-Tiefenbacher U, Sutterlin M, Esserman L, Holtveg HM, Roncadin M, Pigorsch S, Metaxas M, Falzon M, Matthews A, Corica T, Williams NR, Baum M. Targeted intraoperative radiotherapy versus whole breast radiotherapy for breast cancer (TARGIT-A trial): an international, prospective, randomised, non-inferiority phase 3 trial. Lancet. 2010 Jul 10;376(9735):91-102. doi: 10.1016/S0140-6736(10)60837-9. PMID 20570343
- [Background] Veronesi U, Orecchia R, Luini A, Galimberti V, Zurrida S, Intra M, Veronesi P, Arnone P, Leonardi MC, Ciocca M, Lazzari R, Caldarella P, Rotmensz N, Sangalli C, Sances D, Maisonneuve P. Intraoperative radiotherapy during breast conserving surgery: a study on 1,822 cases treated with electrons. Breast Cancer Res Treat. 2010 Nov;124(1):141-51. doi: 10.1007/s10549-010-1115-5. Epub 2010 Aug 15. PMID 20711810
- [Background] Veronesi U, Orecchia R, Maisonneuve P, Viale G, Rotmensz N, Sangalli C, Luini A, Veronesi P, Galimberti V, Zurrida S, Leonardi MC, Lazzari R, Cattani F, Gentilini O, Intra M, Caldarella P, Ballardini B. Intraoperative radiotherapy versus external radiotherapy for early breast cancer (ELIOT): a randomised controlled equivalence trial. Lancet Oncol. 2013 Dec;14(13):1269-77. doi: 10.1016/S1470-2045(13)70497-2. Epub 2013 Nov 11. PMID 24225155
- [Background] Videtic GM, Stephans KL. The role of stereotactic body radiotherapy in the management of non-small cell lung cancer: an emerging standard for the medically inoperable patient? Curr Oncol Rep. 2010 Jul;12(4):235-41. doi: 10.1007/s11912-010-0108-1. PMID 20446066